CLINICAL TRIAL: NCT00266357
Title: MK0928 Phase II Sleep Laboratory Study - Primary Insomnia
Brief Title: Sleep Laboratory Study of MK0928 in Adult Patients With Primary Insomnia (0928-041)(TERMINATED)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0928-041; 2005_107
Record Dates: First submitted 2005-12-14; First posted 2005-12-16 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Primary Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — gaboxadol; Duration of Therapy

INTERVENTIONS:
Drug: MK0928, gaboxadol / Duration of Treatment: 6 days for treatment periods (2 days/dose)
Drug: Placebo / Duration of Treatment: 2 days for screening period

SUMMARY:
A study to evaluate the efficacy, safety and tolerability of MK-0928 in Primary Insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of primary insomnia

Exclusion Criteria:

* Patients with an active psychiatric disorder other than primary insomnia

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50
Dates: Start 2005-11; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Mean of total sleep time over 2 nights.

SECONDARY OUTCOMES:
Mean of other PSG sleep parameters over 2 nights, mean of subjective sleep parameters, and exploratory residual effect.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC